CLINICAL TRIAL: NCT04884620
Title: The COPENHAGEN School Study. Normal Pubertal Development in Youth 2021 and Long-term Disease and Death Risk After Extremely Early Puberty
Brief Title: The 3rd COPENHAGEN Puberty Study
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); European Commission (Other)
Responsible Party: Principal Investigator, Anders Juul, Anders Juul, Rigshospitalet, Denmark, Rigshospitalet, Denmark
Other Study IDs: CopenhagenPuberty3
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Puberty; Puberty, Precocious
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples, serum, white cells, urine, dried blood spots.
  DNA and RNA will be isolated and amplified from collected blood samples and stored. Only specific primers targeted at known SNPs in genes with established or theoretic effects on hormone production, modification or receptor sensitivity or SNP arrays covering common variants (≥1% minor allele frequency, based on allele frequency of the population reference in the current standard, e.g. "The Haplotype Reference Consortium") will be used for genetic analysis. Genetic analysis will not include extensive mapping of the human genome. SNP array data are important at the group level for scientific purposes, but not valid for making clinical judgments on the individual level on the health of the participants. We will not determine any genetic diseases. The participants will not be informed of the results of their individual genetic makeup, only group level information will be available.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-sectional cohort: Healthy children and adolescents from twenty-five selected schools in the metropolitan area
- Longitudinal cohort: Cases with first-time diagnoses of extremely early puberty within the period 1995-2019 in the National Patient Registry and five randomly selected references drawn from the general background population in the Danish Civil registry (CPR) matched on age and sex for each case

SUMMARY:
The COPENHAGEN School Study is a combined cross-sectional and longitudinal study of healthy Danish school children. This study will by clinical examinations and withdrawal of blood samples investigate whether age of pubertal onset is continuing to decline in Denmark over the past 15 years. Furthermore, we will investigate the mechanism driving earlier onset of puberty and the long term health risks of extremely early puberty using Danish registry data

DETAILED DESCRIPTION:
Cross-sectional School study:

All children will be examined once and the following data will be collected:

1. Clinical medical examination of the child consisting of height measurements (standing- and sitting-height), arm-span, weight, fat fold measurements (biceps, triceps, flank, subscapularis), circumference of waist and hip, waist-hip ratio, blood pressure, body fat composition. Puberty development will be assessed by trained and experienced clinical personal according to Tanner criteria. Girls will be investigated for assessment of breast development stage B1-5 (by palpation), pubic hair staging PH1-5, occurrence of axillary hair (Stage 0-2), menarche (yes / no), sweat (yes/no) and acne (yes/no), and boys, their genitalia development stage G1-5, pubic hair stage PH1-6, occurrence of axillary hair (yes/no), acne (yes/no), sweat (yes/no), voice frequency, and voice break (yes/no). The testicular volume assessed by means of Praders orchidometer.
2. Blood sample (35 ml) for measurement of: a) Hormone levels, peptides and growth factors (FSH, LH, estradiol (total/free), progesterone, estrone/estrone sulphate, SHBG, testosterone (total/free), DHEAS, 17-hydroxyprogestrerone, androstenedione, 11-dinhibin B, AMH, INSL3 (only boys), kisspeptin, ghrelin, leptin, IGF-1, IGFBP-3, IGF-related peptides, eoxycortisol, cortisol, cortisone, RANKL, OPG, fibroblast growth factor 23 (FGF23), TSH, T4, free T4, T3, free T3, HbA1C, calcium ion, alkaline phosphatase, PTH, magnesium, phosphate, 25-OH-vitamin D, osteocalcin, prolactin, insulin and lipids (HDL, LDL, TG, Ip(a), cholesterol and lipoproteins), blood metabolites (e.g. amino acids, biogenic amines, acylcarnitines, lyso-phosphatidylcholines, phosphatidylcholines, sphingomyelins and hexose) and proteins (e.g. cytokines, growth factors, kinases, plasma receptors, proteases, protease inhibitors, plasma hormones and structural proteins)); b) Endocrine disrupters (PCBs, dioxins, parabens and phtalates); and c) DNA and RNA
3. Spot urine sample (100 ml) for measurement of FSH, LH, testosterone and endocrine disrupters ( parabens, pthalates, bisphenol A, UV-filters and triclosan)
4. Self-administered electronic questionnaire collecting information on previous growth, illness, living conditions, lifestyle factors, parents' puberty history and current hight and weight.

Biobank Blood and urine samples will be temporary stored during the data collection period until 30th of July 2026. After this date, all unused serum, urine and DNA/RNA not used in the planned analyses will be stored at the established permanent (RegionH, Fælles Fryserfaciliteter) biobank (BIOSEK). The period of storage here is 30 years from the date that the temporary storage is closed.

Prospective Registry-based Cohort study of the Long-term health and death risk after extremely early puberty:

With a follow-up design, we will assess risk of morbidity and mortality amongst cases and referent children. Hazard rations (HRs) will be calculated using Cox regression analyses with stratification using each case and his/her matched referent subjects as a stratum. This ensures that comparisons are adjusted for age and calendar time. Co-variates includes maternal (BMI, smoking, socioeconomic status) during the index pregnancy, also birth weight, length and head circumference of participants. All will be identified in national registries for all persons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adolescents

Exclusion Criteria:

* In case of acute disease, cancer, cancer therapy, or chronic disease (History of malignant disease, chemotherapy or radiation, cystic fibrosis, juvenile rheumatoid arthritis, systemic lupus erythematosus, sickle cell disease, thalassemia, chronic renal disease or known numerical chromosome aberration)
* Non-Caucasian

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cross-sectional population-based puberty study:
  All children and adolescents from 25 selected schools in the metropolitan area were invited to participate in the study
  Longitudinal register-based follow up study of children with precocious puberty:
  All hospital patient records of first-time diagnoses of extremely early puberty within the period 1995-2019 was identified (N=8596) in the National Patient Registry. Five randomly selected persons matched on age and sex for each case of extremely early puberty diagnosis were drawn from the general background population in the Danish Civil registry (CPR) (n=42,980)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2056-12-31 (Estimated)

PRIMARY OUTCOMES:
Pubertal development | Up to an 8 year period
  Pubertal onset according to Tanner criteria:
  * Girls was investigated for assessment of breast development stage B1-5 (by palpation), pubic hair staging PH1-5, occurrence of axillary hair (Stage 0-2), menarche, sweat and acne.
  * Boys was examined in order to assess their genitalia development stage G1-5, pubic hair stage PH1-6, occurrence of axillary hair, acne, sweat, voice break and testicular volume (Praders orchidometer30).
Long-term disease and death risk after extremely early puberty | Up to a 20 year period
  Diagnoses include cancer (prostate and breast), metabolic syndrome, diabetes type 2, cardiovascular disorders (coronary heart disease, heart failure, stroke), and mental health outcomes (depression (major or chronic), anxiety, attempted suicide). Information on the outcomes of interest were extracted from national registers including the National Patient Register, Psychiatric Central Research Registry, National Prescription Registry, Cancer Registry, Causes of Death Registry40 and Medical Birth Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, PhD, DMSc, Principal Investigator — Rigshospitalet, Department of Growth and Reproduction
Locations (1):
- Rigshospitalet, Department of Growth and Reproduction, Copenhagen, Denmark